CLINICAL TRIAL: NCT01325285
Title: The Response of Intraocular Pressure to Systemic Hypercapnia and Hyperoxia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Toronto (Other)
Collaborators: University Health Network, Toronto (Other); Thornhill Research (Unknown)
Responsible Party: Dr. Christopher Hudson, University of Toronto, University of Waterloo, and Toronto Western Research Institute
Other Study IDs: 10-0655
Record Dates: First submitted 2011-02-15; First posted 2011-03-29 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2010-11

CONDITIONS: Intraocular Pressure
Keywords: Intraocular pressure; Hypercapnia; Hyperoxia; Rebreathing circuit
MeSH Terms: conditions — Hypercapnia; Hyperoxia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: RespirAct — Participants will breathe through a mask connected to a sequential rebreathing circuit and gas blender. The following seven gas stages will be targeted for about 10 minutes each:
  1. Baseline, measured in eye A (PETCO2=38mmHg and PETO2=100mmHg)
  2. 10% hypercapnic increase, measured in eye A (PETCO2=42mmHg and PETO2=100mmHg)
  3. 20% hypercapnic increase, measured in eye A (PETCO2=46mmHg and PETO2=100mmHg)
  4. Baseline, measured in both eyes (PETCO2=38mmHg and PETO2=100mmHg)
  5. 250% hyperoxic increase, measured in eye B (PETCO2=38mmHg and PETO2=250mmHg)
  6. 500% hyperoxic increase, measured in eye B (PETCO2=38mmHg and PETO2=500mmHg)
  7. Baseline, measured in eye B (PETCO2=38mmHg and PETO2=100mmHg)
  Other Names: Inhaled gas provocations

SUMMARY:
The purpose of this study is to determine how intraocular pressure responds to changes in the levels of carbon dioxide or oxygen that a healthy individual inspires.

DETAILED DESCRIPTION:
In response to changes in the composition of inhaled gases, blood vessels will dilate or constrict. As a result, hypercapnia or hyperoxia may affect the production and drainage of aqueous humour in the anterior chamber of the eye. The balance between the production and drainage of the aqueous humour determines the intraocular pressure. As this system is hydrodynamic, it is expected that any increase or decrease in the production of aqueous humour due to dilation or constriction of the capillaries within the ciliary body will be compensated by increased or decreased drainage at the trabecular meshwork. Therefore intraocular pressure is not expected to show a response to hypercapnia or hyperoxia, but this supposition needs to be tested in a stably controlled manner of inducing inhaled gas provocations. This study will measure the intraocular pressure at varying levels of hypercapnia and hyperoxia using a sequential rebreathing circuit and automated gas blender. This will allow the precise targeting and stable control of end-tidal partial pressure values of carbon dioxide and oxygen.

In this study, intraocular pressure will be measured at seven different inhaled gas stages. The seven stages are as follows:

1. Baseline, measured in eye A (PETCO2=38mmHg and PETO2=100mmHg)
2. 10% hypercapnic increase, measured in eye A (PETCO2=42mmHg and PETO2=100mmHg)
3. 20% hypercapnic increase, measured in eye A (PETCO2=46mmHg and PETO2=100mmHg)
4. Baseline, measured in both eyes (PETCO2=38mmHg and PETO2=100mmHg)
5. 250% hyperoxic increase, measured in eye B (PETCO2=38mmHg and PETO2=250mmHg)
6. 500% hyperoxic increase, measured in eye B (PETCO2=38mmHg and PETO2=500mmHg)
7. Baseline, measured in eye B (PETCO2=38mmHg and PETO2=100mmHg)

ELIGIBILITY:
Inclusion Criteria:

* Age range 18-30 years old
* Visual acuity of 20/20 or better

Exclusion Criteria:

* Refractive error >±6.00 DS and/or ± 2.00 DC
* History or presence of ocular disease
* Family history of diabetes or glaucoma
* History of intraocular or refractive surgery
* Nursing or pregnant women
* History of clinically diagnosed endocrine disease
* History of vascular disease, cardiovascular disease, or any treated respiratory disorders (seasonal asthma excluded from this so long as subject not taking Rx at the time)
* History of systemic hypertension
* Habitual smoking
* Use of medications that affect blood flow

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy young individuals (age 18-30)
Sampling Method: Non-Probability Sample
Enrollment: 14 (Estimated)
Dates: Start 2011-08; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | Intraocular pressure will be measured during the study visit, ten minutes into each of the seven inhaled gas provocation stages
  Intraocular pressure will be measured using Goldmann applanation tonometry.

SECONDARY OUTCOMES:
Retinal blood flow | Retinal blood flow will be measured during the second (optional) study visit, ten minutes into each of the seven inhaled gas provocation stages
  Retinal blood flow will be measured using the Canon Laser Blood Flowmeter in a subset of participants asked to return for a second visit. This will demonstrate that retinal blood flow behaves as the study claims that it does.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hudson, PhD, Principal Investigator — University of Toronto
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Hosking SL, Harris A, Chung HS, Jonescu-Cuypers CP, Kagemann L, Roff Hilton EJ, Garzozi H. Ocular haemodynamic responses to induced hypercapnia and hyperoxia in glaucoma. Br J Ophthalmol. 2004 Mar;88(3):406-11. doi: 10.1136/bjo.2002.008995. PMID 14977778
- [Background] Slessarev M, Han J, Mardimae A, Prisman E, Preiss D, Volgyesi G, Ansel C, Duffin J, Fisher JA. Prospective targeting and control of end-tidal CO2 and O2 concentrations. J Physiol. 2007 Jun 15;581(Pt 3):1207-19. doi: 10.1113/jphysiol.2007.129395. Epub 2007 Apr 19. PMID 17446225